CLINICAL TRIAL: NCT04184635
Title: Assessment of ECMO in Acute Myocardial Infarction With Non-reversible Cardiogenic Shock to Halt Organ Failure and Reduce Mortality (ANCHOR)
Brief Title: Assessment of ECMO in Acute Myocardial Infarction Cardiogenic Shock
Acronym: ANCHOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P140936; N°ID-RCB : 2019-A00275-52 (Other: ANSM)
Record Dates: First submitted 2019-11-28; First posted 2019-12-03 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Acute Myocardial Infarction; Cardiogenic Shock
Keywords: cardiogenic shock; VA-ECMO; STEMI; NSTEMI; Intraortic balloon pump
MeSH Terms: conditions — Shock, Cardiogenic; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: A multicenter, prospective, randomized, comparative open trial will be conducted on two parallel groups of patients with AMI complicated by cardiogenic shock.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental ECMO + IABP Arm (Experimental): VA-ECMO will be instituted percutaneously under echo guidance via the femoral route as soon as possible.
  An IABP will be systematically inserted in the contralateral femoral artery (unless technically not possible).
  Interventions: Device: VA-ECMO
- Control Conventional Treatment Arm (No Intervention): Standard management of cardiogenic shock due to myocardial infarction according to the current ESC guidelines. It is not recommended to use IABP support and no other TCS device (e.g., ECMO, Impella, Thoratec PHP, TandemHeart) will be permitted in the control group.

INTERVENTIONS:
Device: VA-ECMO — * The ECMO device will be the CardioHelp (MAQUET, GETINGE, Orléans, France) using the veno-arterial setting and percutaneous femoro-femoral cannulation with MAQUET GETINGE HLS cannulae.
  * Intraortic balloon pump will be MEGA 50 cc or 40cc, (MAQUET, GETINGE, Orléans, France).
  Arms: Experimental ECMO + IABP Arm

SUMMARY:
Data from case series and large retrospective trials suggest that the early treatment of cardiogenic shock AMI patients with the association of VA-ECMO and IABP may significantly decrease mortality, which is still unacceptably high nowadays (40-50% at 30 days).

An important benefit for the patients randomized to the ECMO arm is expected and the risk-to-benefit ratio is expected to be in favor of the experimental treatment arm.

DETAILED DESCRIPTION:
Scientific background

- Venoarterial extracorporeal membrane oxygenation (VA-ECMO) is used more and more frequently in patients with acute myocardial infarction (AMI) and refractory cardiogenic shock despite the absence of high level scientific evidence to recommend the use of temporary circulatory support devices (TCS) in this setting.TCS support may also benefit to cardiogenic shock patients not initially refractory to conventional medical management since their mortality exceeds 40% and most of deaths are due to the development of refractory cardiogenic shock and multiple organ failure.

The ANCHOR trial is therefore designed to test the hypothesis that VA-ECMO support associated with IABP results in improved outcomes in comparison with optimal medical treatment alone in patients with AMI and cardiogenic shock. An ethical rescue option to VA-ECMO will however be provided to control patients with cardiogenic shock refractory to conventional medical treatment since recent data suggested survival up-to 50% with ECMO support in this setting.

Main objective - To determine if early VA-ECMO combined with IABP support and optimal medical treatment would improve the outcomes of patients with acute myocardial infarction complicated by cardiogenic shock as compared with optimal medical treatment alone.

Scope of the study

- Patients satisfying all of the Inclusion and Exclusion Criteria will be classified as 'Eligible'. Consent to research will be obtained from a close relative or surrogate for all eligible patients prior to randomization.

Should such a person be absent, eligible patients will be randomized according to the specifications of emergency consent and the patient will be asked to give his/her consent for the continuation of the trial when his/her condition will allow.

Randomization will be possible in centers with robust experience in the management of AMI and cardiogenic shock but no on-site ECMO capability providing that an ECMO retrieval team from the nearest ECMO center can establish ECMO no later than 2 hours after randomization.

Before randomization, physicians at the non-ECMO center will check that the ECMO team is immediately available and that an ICU/CCU bed is available at the ECMO center. Thereafter, if the patient is randomized to the ECMO arm, the mobile ECMO retrieval team will travel to the center, initiate VA-ECMO and will rapidly transfer the patient on VA-ECMO to the ECMO center.

Description of experimental ECMO + IABP Arm

* Protocolized conventional management of cardiogenic shock
* VA-ECMO will be started as soon as possible
* For patients randomized at non-ECMO centers, a mobile ECMO team will initiate ECMO at the non-ECMO center and transport the patient to the ECMO center immediately
* IABP inserted in the contralateral femoral artery (unless technically not possible)
* ECMO management according to protocol
* ECMO weaning according to protocol

Description of conventional treatment Arm

* Protocolized conventional management of cardiogenic shock
* IABP not recommended. No other TCS device (e.g., ECMO, Impella, Thoratec PHP, TandemHeart) permitted
* Rescue VA-ECMO only if one of 1 or 2 or 3 applies:
* 1. Refractory cardiogenic shock defined as

  1. Cardiac index <1.2 l/min/m² or VTI <6 cm AND
  2. Assessment and correction of hypovolemia AND
  3. (dobutamine ≥15 microg/kg/min + norepinephrine ≥1.5 microg/kg/min) OR epinephrine ≥ 0.75 microg/kg/min
  4. Serum lactate >5 mmol/L or serum lactate increased >50% in the last 6 hours
* 2. Uncontrolled lethal arrhythmia despite K >4.5 mmol/l AND Mg >1.0 mmol/l AND Intubation and mechanical ventilation with deep sedation AND IV Loading of amiodarone AND IV xylocaine
* 3. Refractory cardiac arrest

Mandatory validation of rescue VA-ECMO by an independent adjudicator.

ELIGIBILITY:
Inclusion Criteria:

* Cardiogenic shock complicating acute myocardial infarction (STEMI or NSTEMI)
* Revascularization by PCI for acute myocardial infarction has been performed or is planned in the following 60 minutes
* Systolic blood pressure <90 mmHg for >30 min or catecholamine support required to maintain systolic blood pressure >90 mmHg
* Signs of pulmonary congestion
* Signs of impaired organ perfusion with at least one of the following:

Altered mental status OR cold, clammy skin and extremities OR oliguria with urine output <30 ml/h OR serum lactate >2.0 mmol/l

Exclusion Criteria:

* Age <18 years
* Pregnancy
* Onset of shock >24 Hours
* Shock of other cause (hypovolemic, anaphylactic or vagal shock)
* Shock due to massive pulmonary embolism
* Resuscitation >30 minutes
* No intrinsic heart activity
* Patient moribund on the day of randomization or SAPS II >90
* Surgical revascularization for AMI (CABG) planned or already performed prior to randomization
* Cerebral deficit with fixed dilated pupils or Irreversible neurological pathology
* Mechanical infarction complication (massive mitral regurgitation, pericardium drainage required, septal ventricular defect)
* Severe peripheral artery disease or previous aortic or ilio-femoral surgery precluding ECMO and IABP insertion
* Aortic regurgitation > II
* Other severe concomitant disease with limited life expectancy < 1 year
* Proven heparin-induced thrombocytopenia
* ECMO device not immediately available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-10-14 (Actual); Primary Completion 2026-10-14 (Estimated); Study Completion 2027-10-14 (Estimated)

PRIMARY OUTCOMES:
Treatment failure at Day 30 | At day 30
  Death in the ECMO group and death OR rescue ECMO in the control group

SECONDARY OUTCOMES:
Mortality at Day 30 | At day 30
  All-cause mortality at day 30
Major Adverse Cardiovascular Events | At day 30
  Major Adverse Cardiovascular Events are defined as death, stroke (any new neurological symptoms in association with signs of ischemia or hemorrhage in a cranial CT or MRI), recurrent myocardial infarction, need for repeat revascularization (PCI and/or CABG), renal replacement therapy, re-hospitalization for heart failure, escalation to permanent left ventricular assist device (LVAD) or total artificial heart, cardiac transplant.
Stroke | At day 30
  Any new neurological symptoms in association with signs of ischemia or hemorrhage in a cranial CT or MRI
Recurrent myocardial infarction | At day 30
  Recurrent myocardial infarction
Need for repeat revascularization with PCI and/or CABG | At day 30
  Need for repeat revascularization (PCI and/or CABG)
Need for renal replacement therapy | At day 30
  Need for renal replacement therapy
Re-hospitalization for heart failure | At day 30
  re-hospitalization for heart failure
Escalation to LVAD or total artificial heart | At day 30
  Escalation to permanent left ventricular assist device or total artificial heart
Cardiac transplantation | At day 30
  Cardiac transplantation
Major bleeding | At day 30
  Major bleeding (TIMI definition): Any intracranial bleeding (excluding microhemorrhages <10 mm evident only on gradient-echo MRI) OR Clinically overt signs of hemorrhage associated with a drop in hemoglobin of ≥5 g/dL or a ≥15% absolute decrease in hematocrit OR Fatal bleeding (bleeding that directly results in death within 7 d)
Red blood cells transfused | At day 30
  Number of packed red blood cells transfused
Serum lactate | At day 30
  Time to serum lactate normalization
Number of days alive without organ failure at day 30 | At day 30
  Number of days alive without organ failure(s) defined with the SOFA score, catecholamine support, mechanical ventilation and renal replacement therapy
Durations of ICU stay and hospitalization | At day 30
  Durations of ICU stay and of hospitalization
LV function | At day 30
  LV function assessed with Doppler echocardiography or magnetic resonance imaging
NYHA/INTERMACS status | At day 30
  NYHA/INTERMACS status
ECMO-related complications | At day 30
  ECMO-related complications (infection at VA-ECMO cannulation sites requiring antibiotics, hemorrhage, limb ischemia requiring surgery, cannula or circuit thrombosis, overt pulmonary edema, thrombocytopenia, gaseous emboli and hemolysis).
Treatment failure at one year | At one year
  Treatment failure defined as death (all-cause) in the ECMO group and death (all-cause) OR rescue ECMO in the control group.
Mortality at one year | At one year
  All-cause mortality
Major Adverse Cardiovascular at one year | At one year
  MACE, Major Adverse Cardiovascular Events are defined as death, stroke (any new neurological symptoms in association with signs of ischemia or hemorrhage in a cranial CT or MRI), recurrent myocardial infarction, need for repeat revascularization (PCI and/or CABG), renal replacement therapy, re-hospitalization for heart failure, escalation to permanent left ventricular assist device (LVAD) or total artificial heart, cardiac transplant.
Stroke at one year | At one year
  Stroke (any new neurological symptoms in association with signs of ischemia or hemorrhage in a cranial CT or MRI),
Recurrent myocardial infarction at one year | At one year
  Recurrent myocardial infarction between randomization and one year
PCI and/or CABG at one year | At one year
  Repeat revascularization (PCI and/or CABG) between randomization and one year
Renal replacement therapy at one year | At one year
  Need for renal replacement therapy between randomization and one year
Re-hospitalization for heart failure | At one year
  Re-hospitalization for heart failure between randomization and one year
LVAD at one year | At one year
  Escalation to permanent left ventricular assist device (LVAD) or total artificial heart
Cardiac transplant at one year | At one year
  Cardiac transplantation
Major bleeding at one year | At one year
  Major bleeding (TIMI definition): Any intracranial bleeding (excluding microhemorrhages <10 mm evident only on gradient-echo MRI) OR Clinically overt signs of hemorrhage associated with a drop in hemoglobin of ≥5 g/dL or a ≥15% absolute decrease in hematocrit OR Fatal bleeding (bleeding that directly results in death within 7 d)
NYHA/INTERMACS status at one year | At one year
  NYHA/INTERMACS status
Returned to work at one year | At one year
  Rate of patients who returned to work if previously active
LV ejection fraction at one year | At one year
  Latest LV ejection fraction
Short Form 36 (SF-36) questionnaire at one year | At one year
  Quality of life assessed using the Short Form 36 (SF-36) Health Survey questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Alain COMBES, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire Pitié-Salpêtrière Paris
Locations (1):
- Hôpital Pitié Salpétrière, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thiele H, Akin I, Sandri M, Fuernau G, de Waha S, Meyer-Saraei R, Nordbeck P, Geisler T, Landmesser U, Skurk C, Fach A, Lapp H, Piek JJ, Noc M, Goslar T, Felix SB, Maier LS, Stepinska J, Oldroyd K, Serpytis P, Montalescot G, Barthelemy O, Huber K, Windecker S, Savonitto S, Torremante P, Vrints C, Schneider S, Desch S, Zeymer U; CULPRIT-SHOCK Investigators. PCI Strategies in Patients with Acute Myocardial Infarction and Cardiogenic Shock. N Engl J Med. 2017 Dec 21;377(25):2419-2432. doi: 10.1056/NEJMoa1710261. Epub 2017 Oct 30. PMID 29083953
- [Background] Authors/Task Force members; Windecker S, Kolh P, Alfonso F, Collet JP, Cremer J, Falk V, Filippatos G, Hamm C, Head SJ, Juni P, Kappetein AP, Kastrati A, Knuuti J, Landmesser U, Laufer G, Neumann FJ, Richter DJ, Schauerte P, Sousa Uva M, Stefanini GG, Taggart DP, Torracca L, Valgimigli M, Wijns W, Witkowski A. 2014 ESC/EACTS Guidelines on myocardial revascularization: The Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS)Developed with the special contribution of the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eur Heart J. 2014 Oct 1;35(37):2541-619. doi: 10.1093/eurheartj/ehu278. Epub 2014 Aug 29. No abstract available. PMID 25173339
- [Background] Thiele H, Akin I, Sandri M, de Waha-Thiele S, Meyer-Saraei R, Fuernau G, Eitel I, Nordbeck P, Geisler T, Landmesser U, Skurk C, Fach A, Jobs A, Lapp H, Piek JJ, Noc M, Goslar T, Felix SB, Maier LS, Stepinska J, Oldroyd K, Serpytis P, Montalescot G, Barthelemy O, Huber K, Windecker S, Hunziker L, Savonitto S, Torremante P, Vrints C, Schneider S, Zeymer U, Desch S; CULPRIT-SHOCK Investigators. One-Year Outcomes after PCI Strategies in Cardiogenic Shock. N Engl J Med. 2018 Nov 1;379(18):1699-1710. doi: 10.1056/NEJMoa1808788. Epub 2018 Aug 25. PMID 30145971
- [Background] Overtchouk P, Pascal J, Lebreton G, Hulot JS, Luyt CE, Combes A, Kerneis M, Silvain J, Barthelemy O, Leprince P, Brechot N, Montalescot G, Collet JP. Outcome after revascularisation of acute myocardial infarction with cardiogenic shock on extracorporeal life support. EuroIntervention. 2018 Apr 6;13(18):e2160-e2168. doi: 10.4244/EIJ-D-17-01014. PMID 29400656
- [Background] Muller G, Flecher E, Lebreton G, Luyt CE, Trouillet JL, Brechot N, Schmidt M, Mastroianni C, Chastre J, Leprince P, Anselmi A, Combes A. The ENCOURAGE mortality risk score and analysis of long-term outcomes after VA-ECMO for acute myocardial infarction with cardiogenic shock. Intensive Care Med. 2016 Mar;42(3):370-378. doi: 10.1007/s00134-016-4223-9. Epub 2016 Jan 29. PMID 26825953